CLINICAL TRIAL: NCT05853523
Title: The Desensitizing Treatment Effects of the Laser and Ozone on Dentin Hypersensitivity: In-vivo Comparison
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Maurizio D'Amario, Dott. Maurizio D'Amario, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CONS 01_21
Record Dates: First submitted 2023-04-29; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: Split Mouth: all patients involved received both treatments randomly assigned to either the right or left halves of the dentition.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gas ozone group (Experimental): Participant received 32 g/m3 of gas ozone for 30 second.
  Interventions: Combination Product: Gas ozone
- Diode laser group (Experimental): Participant received an application of desensitized gel, fluoride and potassium nitrate gel , and a first step of an irradiation with diode laser for 20 second of interval, 808 wavelength, and power incrementation, from 0,2 till 0,6 W, not in contact. Then the second step of irradiation for 30 second in contact with dentine surface, 808 wavelength, and power incrementation, from 0,2 till 0,6 W. Then the surface was rinsed, and the irradiation applied for a third time again without the gel as the second step.
  Interventions: Combination Product: Diode laser and desensitized gel

INTERVENTIONS:
Combination Product: Gas ozone — The application of ozone was performed with the HealOzone System X4 (HealOzon, Kavo, Germany). The dentist adapted the silicon cup stricken on the cervical surface of the teeth. The pumping system created the vacuum and the machine applied high dosage of ozone, equal to 32 g/m3, for 30 second.
  Arms: Gas ozone group
Combination Product: Diode laser and desensitized gel — The dentist applied desensitized gel (JW-Desensitizing Gel, Heydent Gmbh, Germany) directly on the cervical zone of the teeth. Subsequently the irradiation was performed with Wiser III (Wiser, Doctor Smile, Italy) in the desensitizing assisted mode (preprogramed protocol). The protocol provides consecutively steps (not in contact) with 20 second of interval, 808 wavelength, and power incrementation, from 0,2 till 0,6 W. radiating the entire desensitize surface second using the "black tip" (400 micron). The procedure continued maintaining the tip of the laser on contact with the dentine surface making movement of lawn mowing (brushing technique) for 30 second. Then the surface was rinsed, and the irradiation applied again without the gel.
  Arms: Diode laser group

SUMMARY:
The goal of this split mouth clinical trial is to compare clinical efficacy of diode laser and gas ozone in the treatment of dentine hypersensitivity (DHS) of non-carious-cervical lesion. The main questions it aims to answer are:

* gas ozone affects dentine hypersensitivity?
* diode laser affects dentine hypersensitivity? Participants, affected of DHS , were treated with gas ozone and diode laser.The pain severity was quantified according to the Visual Analogue Scale (VAS) before and after the treatmens.

ELIGIBILITY:
Inclusion Criteria:

* Stimulated dentine hypersensitivity greater than 6 on visual analogue scale (VAS)
* DHS affected two teeth, not contiguous, of different mouth semiarch.

Exclusion Criteria:

* Periodontal surgery in the last 3 month
* Use of desensitizing paste in the last 3 month
* Pregnant or breastfeeding state
* Teeth with caries, reconstructions, pulpits congenital anomalies, fracture, and occlusal interferences.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-27 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-08-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain on the 10-point Visual Analogue Scale (VAS) immediately after treatment | 5 minutes
  Two stimuli were adopted to assess the degree of dentine hypersensitivities: evaporative test and tactile test. For the evaporative test, the teeth were trigged by a single operator, experienced, and trained, with a jet of air at a pressure of 45-60 psi at a distance of 2 mm from the buccal surface for 35 s. For the tactile test, the pain was triggered using a probe gently touched the dentine exposed in mesiodistal direction. The patient quantified the pain with the visual analogue scale (VAS) giving a value in the range from 1 (minimum pain) to 10 (maximum pain). The highest value of the pain stimulated by the two methods was registered.
Pain on the 10-point Visual Analogue Scale (VAS) at 3 months from treatment | 3 months
  Two stimuli were adopted to assess the degree of dentine hypersensitivities: evaporative test and tactile test. For the evaporative test, the teeth were trigged by a single operator, experienced, and trained, with a jet of air at a pressure of 45-60 psi at a distance of 2 mm from the buccal surface for 35 s. For the tactile test, the pain was triggered using a probe gently touched the dentine exposed in mesiodistal direction. The patient quantified the pain with the visual analogue scale (VAS) giving a value in the range from 1 (minimum pain) to 10 (maximum pain). The highest value of the pain stimulated by the two methods was registered.
Pain on the 10-point Visual Analogue Scale (VAS) at 6 months from treatment | 6 months
  Two stimuli were adopted to assess the degree of dentine hypersensitivities: evaporative test and tactile test. For the evaporative test, the teeth were trigged by a single operator, experienced, and trained, with a jet of air at a pressure of 45-60 psi at a distance of 2 mm from the buccal surface for 35 s. For the tactile test, the pain was triggered using a probe gently touched the dentine exposed in mesiodistal direction. The patient quantified the pain with the visual analogue scale (VAS) giving a value in the range from 1 (minimum pain) to 10 (maximum pain). The highest value of the pain stimulated by the two methods was registered.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio D'Amario, Principal Investigator — University of L'Aquila
Locations (1):
- University of L'Aquila, L’Aquila, AQ, Italy

REFERENCES:
- [Background] Holland GR, Narhi MN, Addy M, Gangarosa L, Orchardson R. Guidelines for the design and conduct of clinical trials on dentine hypersensitivity. J Clin Periodontol. 1997 Nov;24(11):808-13. doi: 10.1111/j.1600-051x.1997.tb01194.x. PMID 9402502